CLINICAL TRIAL: NCT01244477
Title: Neuroimaging the Impact of Treatment on Neural Substrates of Trust in PTSD
Brief Title: Neuroimaging the Impact of Treatment on Neural Substrates of Trust in Post-Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B7760-P
Record Dates: First submitted 2010-11-17; First posted 2010-11-19 (Estimated); Results first posted 2014-12-02 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Stress Disorders, Post Traumatic; Trust
Keywords: Stress Disorders, Post Traumatic; Trust; functional Magnetic Resonance Imaging (fMRI)
MeSH Terms: conditions — Combat Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CPT-C (Experimental): Participants in group CPT-C
  Interventions: Behavioral: Group CPT-C
- Treatment-as-Usual (No Intervention): Participants randomly assigned to the Waitlist Control Group (who will participate in CPT-C after 12 weeks).

INTERVENTIONS:
Behavioral: Group CPT-C — Participants will be randomly assigned to participate in CPT-C or a 12 week waitlist control group. Waitlist control subjects will participate in CPT-C after the 12 weeks.
  Arms: CPT-C

SUMMARY:
Traumatic experiences can have a profound negative effect on the lives and well-being of both the people who experience them and their loved ones. For those who experience post-traumatic stress disorder (PTSD), their interpersonal difficulties and social support further impact the success of treatment such that interpersonal difficulties are associated with mistrust and predict poor treatment outcome. In this proposal, the investigators use functional neuroimaging to understand the neurobiology of trust and mistrust in people with PTSD and to learn more about how successful treatment can improve trust and social functioning.

DETAILED DESCRIPTION:
Substantial recent data highlight the role of social functioning as a primary moderator of therapeutic response in individuals with post-traumatic stress disorder (PTSD) such that interpersonal difficulties and mistrust significantly and negatively impact treatment efficacy (Forbes et al., 2003; Forbes et al., 2005; Forbes et al., 2008). In addition, ample evidence suggests that psychotherapy improves the social and interpersonal lives of psychotherapy clients through improving clients' abilities to regulate their emotions and reduce social isolation (Yalom & Leszcz, 2005; Foy et al., 2000). While considerable research has been dedicated to exploring the neurobiology of emotional dysregulation associated with PTSD (Rauch, Shin, & Phelps, 2006; Etkin & Wager, 2007), and increasing data suggest that diverse psychotherapies affect neural functioning (Beauregard 2007), very little is understood about the neurobehavioral pathology underlying the debilitating interpersonal difficulties in PTSD, or the neurobiological mechanisms accompanying the improvements in social functioning that occur with efficacious therapy.

Thus, the broad goals of this project are two-fold. First, the investigators seek to examine the neural substrates associated with interpersonal dysfunction in PTSD using a social exchange game previously developed to assess interpersonal trust and cooperation in healthy (King-Casas et al., 2005) and psychiatric groups (Chiu et al., 2008; King-Casas et al., 2008). Second, the investigators seek to examine changes in neurobehavioral substrates of social functioning following treatment for Veterans with PTSD. Specifically, the investigators propose to use functional magnetic resonance imaging (fMRI) and behavior within a well-characterized Trust Game to examine the neural substrates associated with interpersonal trust and cooperation in Veterans with PTSD prior to and following empirically supported psychotherapy cognitive processing therapy (CPT) for PTSD.

Thus, the broad goals of this project are two-fold. First, the investigators seek to examine the neural substrates associated with interpersonal dysfunction in PTSD using a social exchange game previously developed to assess interpersonal trust and cooperation in healthy (King-Casas et al., 2005) and psychiatric groups (Chiu et al., 2008; King-Casas et al., 2008). Second, the investigators seek to examine changes in neurobehavioral substrates of social functioning following treatment for veterans with PTSD. Specifically, the investigators propose to use functional magnetic resonance imaging (fMRI) and behavior within a well-characterized Trust Game to examine the neural substrates associated with interpersonal trust and cooperation in veterans with PTSD prior to and following empirically supported psychotherapy cognitive processing therapy (CPT) for PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for PTSD on the Clinician Administered PTSD Scale (CAPS)
* Priority will be given to Veterans aged 18-50 who have had an onset of symptoms in the past 10 years and are Veterans of Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF)
* Have been referred for placement in CPT treatment by a clinician in the Trauma Recovery Program at the Michael E DeBakey VA Medical Center (MEDVAMC) or an eligible Veteran who contacts study staff.
* Are able to see the computer display clearly with or without magnetic Resonance imaging (MRI)-compatible corrective lenses
* Are free from current non-psychiatric medical problems impacting cognitive functioning.
* Are cleared to participate by a treating MEDVAMC clinician
* Are able to participate in functional MRI (fMRI)

Exclusion Criteria:

* Meet Diagnostic and Statistical Manual-IV (DSM-IV)criteria for drug or alcohol abuse in the past 30 days
* History of moderate to severe traumatic brain injury based on any of the following:

  * (i) Glasgow Coma Score < 13
  * (ii)alteration of consciousness > 24 hours; loss of consciousness,30 minutes
* Presence of contraindications to MRI, including but not limited to:

  * claustrophobia
  * pacemaker
  * metal in eyes
  * other implants
* Current neurological or general medical conditions known to impact cognitive and/or emotional functioning, including but limited to:

  * epilepsy
  * Parkinson's disease
  * Huntington's disease
  * Alzheimer's disease
  * stroke
  * chemotherapy for cancer
* Acute psychological instability as assessed by a Michael E DeBakey VA Medical Center (MEDVAMC) clinician or study staff
* Concurrent diagnosis of:

  * schizophrenia
  * schizoaffective disorder
  * delusional disorder
  * organic psychosis
  * and subjects taking antipsychotic medication

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2011-05-16 (Actual); Primary Completion 2013-05-31 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wright Williams, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CPT-C: Group Cognitive Processing Therapy-C (CPT-C): Participants who chose to participate in a 12-week CPT-C treatment group.
- Treatment-as-Usual: Participants who chose to participate in a 12-week treatment as usual group and offered CPT-C group treatment after 12 weeks.
Period: Overall Study
Arm/Group | CPT-C | Treatment-as-Usual
Started | 38 | 23
Completed | 18 | 20
Not Completed | 20 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CPT-C | Treatment-as-Usual | Total
Number analyzed (Participants) | 38 | 23 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 23 | 61
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 31 | 19 | 50
Race/Ethnicity, Customized [Number; unit: participants]
  Black/African American | 13 | 5 | 18
  Hispanic or Latino | 6 | 5 | 11
  Mixed Race | 4 | 1 | 5
  Caucasian or White | 15 | 12 | 27

OUTCOME MEASURES:

1. Primary Outcome: Continuous Whole Brain Imaging With Standard Imaging Parameters for Each Functional Magnetic Resonance Imaging (fMRI) Scan
Time Frame: Pre & post a 12 week treatment group
Population: Neural data is not analyzable - scanner technicians changed the parameters of the task fMRI on an unpredictable basis. Project staff and data no longer available.
Groups:
- Arm 1: CPT-C Group: Participants in group CPT-C
  Group CPT-C: Participants will be randomly assigned to participate in CPT-C or a 12 week waitlist control group. Waitlist control subjects will participate in CPT-C after the 12 weeks.
- Arm 2: Waitlist Control Group: Participants randomly assigned to the Waitlist Control Group (who will participate in CPT-C after 12 weeks).
Arm/Group | Arm 1: CPT-C Group | Arm 2: Waitlist Control Group
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: The Clinician Administered PTSD Scale (CAPS)
Description: The CAPS is considered the gold standard measure of PTSD symptoms. CAPS scores are the sum of 17 questions. Each is question is scored from 0 (best possible outcome) to 8 (worst possible outcome). The lowest possible CAPS score is a 0, indicating no PTSD symptoms reported. The highest possible CAPS score is a 136, indicating the most PTSD symptoms reported.
Time Frame: Pre & post a 12 week treatment group
Population: We limited this arm to 18 subjects who completed 9+ out of 12 treatment sessions.
Measure: Mean (Standard Deviation); unit: CAPS Scores
Groups:
- CPT-C: Participants in group CPT-C
  Group CPT-C: Participants who chose to participate in a 12-week CPT-C treatment group.
Arm/Group | CPT-C | Treatment-as-Usual
Number analyzed (Participants) | 18 | 20
CAPS Scores
  Pre-Therapy or before 12 weeks | 79.3 (18.6) | 66.3 (26.2)
  Post-Therapy or after 12 weeks | 70.3 (24.1) | 69.5 (22.8)

3. Secondary Outcome: Behavioral Expression of Trust on the Trust Game
Description: The Investment Ratio (IR) is the amount subjects were willing to invest in a social partner. It is considered a measure of interpersonal trust, and co-operation. It is a ratio ranging from 0 (indicating no willingness to trust a social partner) to 1.0 (willing to totally trust a social partner). It consists of the percentage of total points the subject was willing to invest in a social partner divided by the total points they received for all ten rounds of the trust game. Higher ratio's indicate more trust.
Time Frame: Pre & post a 12 week treatment group
Population: Veterans with PTSD under 50 years of age
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | CPT-C | Treatment-as-Usual
Number analyzed (Participants) | 18 | 20
Ratio
  Pre-Treatment Investment Ratio | .31 (.17) | .34 (.23)
  Post-Treatment Investment Ratio | .37 (.27) | .28 (.25)

4. Secondary Outcome: PTSD Checklist (PCL)
Description: An instrument measuring a participants self-reported level of PTSD symptoms. PCL scores are the sum of 17 questions. Each is question is scored from 1 (best possible outcome) to 5 (worst possible outcome). The lowest possible PCL score is a 17, indicating no troublesome PTSD symptoms reported. The highest possible PCL score is a 85, indicating the worst degree of PTSD symptoms reported.
Time Frame: Administered each week at weekly group sessions or pre-post treatment as usual
Population: Veterans under 50 years of age diagnosed with PTSD
Measure: Mean (Standard Deviation); unit: PCL Scores
Arm/Group | CPT-C | Treatment-as-Usual
Number analyzed (Participants) | 18 | 19
PCL Scores
  Pre-Treatment PCL-M Scores | 65.33 (11.0) | 56.83 (17.1)
  Post-Treatment PCL-M Scores | 58.37 (13.48) | 59.53 (11.88)

ADVERSE EVENTS:
Arm/Group | CPT-C | Treatment-as-Usual
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/23
Other Adverse Events (participants affected / at risk) | 0/38 | 0/23

LIMITATIONS AND CAVEATS:
This is a pilot study based on a small sample of Veterans with PTSD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes